CLINICAL TRIAL: NCT05579704
Title: Digital Intervention for Behaviour Change and Chronic Disease Prevention
Acronym: DIRECTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00121051
Record Dates: First submitted 2022-10-03; First posted 2022-10-14 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based wellness platform (Active Comparator): Participants will receive access to a web-based wellness platform focused on nutrition, physical activity, and mindfulness. Interactions with the platform will be fully self-guided (without weekly group video conferencing sessions healthcare professionals and peers).
  Interventions: Behavioral: Web-based wellness platform
- Web-based wellness platform with healthcare professional-facilitated online support (Experimental): Participants will receive access to a web-based wellness platform focused on nutrition, physical activity, and mindfulness. In addition to the platform access, participants will take part in weekly group video conferencing sessions with various healthcare professionals (registered dietitian, mental health therapist, and exercise professional). The sessions will occur once per week for 1 hour each. The group sessions will contain cohorts of approximately 10 individuals.
  Interventions: Behavioral: Web-based wellness platform; Behavioral: Healthcare professional-facilitated online support group

INTERVENTIONS:
Behavioral: Web-based wellness platform — A web-based wellness platform is based on preventive self-care and contains tools to monitor nutrition, physical activity, and mental wellbeing.
Behavioral: Healthcare professional-facilitated online support group — Participants will take part in weekly group video conferencing sessions with various health professionals (registered dietitian, mental health therapist, and exercise professional). The sessions will occur once per week for 1 hour each. The group sessions will contain cohorts of approximately 10 individuals.
  Arms: Web-based wellness platform with healthcare professional-facilitated online support

SUMMARY:
Body weight, diet quality, physical activity, stress, sleep and alcohol use will be evaluated in a sample of 180 Albertans with excess body weight. Participants will be randomized into the following two groups; active control arm (access to a preventative self-care web-based platform for 16 weeks) vs. intervention arm (access to a preventative self-care web-based platform for 16 weeks plus health professional guidance and supervision).

DETAILED DESCRIPTION:
Excess body weight, poor diet, physical inactivity, alcohol consumption, stress, and sleep deprivation/disruption are modifiable risk factors associated with chronic diseases, such as cancer. While most Canadians may be aware that these play a role in chronic disease prevention, individualized tools are needed to foster sustainable, long-term habits.

Digital health solutions have become commonplace in self-care. They offer an opportunity to reach a large number of individuals with personalized programs to improve health and lower the risk of developing chronic disease. Many digital applications are available for individuals to monitor their diet, activity and weight; however, few have been validated and are based on scientific evidence.

Recently, a Canadian web-based platform centered on preventive self-care became available. This platform was created by health care professionals and encompasses three key pillars of health: nutrition, physical activity, and mindfulness. The effectiveness of this web-based wellness platform will be evaluated in people living with excess body weight to improve six chronic disease risk factors: body weight, diet quality, physical activity, alcohol intake, stress, and sleep habits. A fully self-guided approach (active control, Arm 1) will be compared to an approach guided by a healthcare professional (Arm 2) and compare risk factors pre- and post-intervention. Investigators hypothesize that both approaches will improve modifiable risk factors, but participants guided by a healthcare professional will have greater improvements. Qualitatively, the experiences of immigrants using the platform will be explored.

Participants will use the web-based platform for 16 weeks. Our primary outcome is between-group difference in weight loss. Secondary outcomes include improvements in dietary intake, physical activity and sleep quality, and decrease in alcohol intake and stress. To assess the primary and one of the secondary outcomes (physical activity), a smart scale and a wearable device will be used. Wearable devices are widely used and an effective approach to body weight reduction. Additionally, immigrants' experiences and perspectives of participating in this study will be explored using semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Albertans with excess body weight (BMI 30-35 kg/m2)
* Individuals who are seeking weight loss as screened by the S-Weight Questionnaire
* Ages 40-65 years of age, any sex/gender
* Able to safely exercise as screened by the 2022 Physical Activity Readiness Questionnaire (PAR-Q+)
* Must have a cell phone with internet access and Bluetooth capabilities
* Able to participate in video conferencing on evenings and/or weekends
* Willing to wear a Fitbit activity monitor on the wrist for 16 weeks.
* Able to speak, read and understand English

Exclusion Criteria:

* Participating in intensive lifestyle interventions, structured exercise programming (> 3hrs of vigorous physical activity per week) or structured diet programming
* Taking any medication or supplements that may alter energy metabolism, body weight and composition, as evaluated by study investigators;
* Chronic conditions in which weight loss is not indicated or controversial. Significant medical self-reported comorbidities, including uncontrolled metabolic disorders (e.g., cancer, thyroid, stroke, kidney, liver, respiratory, heart disease, type 1 or uncontrolled type 2 diabetes)
* Self-reported eating disorders, untreated depression, anxiety or other mood disorders
* Weight loss greater than 25 lbs (11 kg) in the past 6 months
* Previous bariatric surgery
* Active substance abuse (alcohol, cannabis, illicit drugs, prescription drugs)
* Unable to adhere to the study protocol

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Change in body weight. | Baseline to Week 16.
  Body weight changes will be measured using Bluetooth enabled smart scales (Fitbit Aria scale) for daily tracking of body weight.

SECONDARY OUTCOMES:
Change in diet quality. | Baseline to Week 16.
  Diet quality changes will be assessed using the Canadian version of the Healthy Eating Index (HEI) measured using the Automated Self-Administered 24-h Dietary Assessment Tool (ASA 24).
Change in self-reported physical activity. | Baseline to Week 16.
  Self-reported physical activity will be assessed using the Godin-Shephard Leisure Time Physical Activity Questionnaire (GLTEQ). Scored as a range from 0 to 24+, where <14 indicates sedentary, 14-23 indicates moderately active and >24 indicates active.
Change in measured step counts. | Baseline to Week 16.
  Physical activity changes will be measured using a wrist-worn wearable activity monitor (Fitbit Inspire 2) to track step counts.
Change in physical activity. | Baseline to Week 16.
  Physical activity changes will be measured using a wrist-worn wearable activity monitor (Fitbit Inspire 2) to track active minutes.
Change in self-reported stress. | Baseline to Week 16.
  Self-reported stress will be assessed using the Perceived Stress Scale (PSS). Scored as a range from 0 to 40, where <14 indicates low stress, 14-26 indicates moderate stress and >26 indicates high perceived stress.
Change in self-reported sleep quality. | Baseline to Week 16.
  Self-reported sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). Scored as a range from 0 to 21, where a higher score indicates worse sleep quality.
Change in self-reported alcohol use. | Baseline to Week 16.
  Self-reported alcohol use will be assessed using the Alcohol Use Disorders Identification Test (AUDIT). Scored as a range from 0 to 40, where a score of 0 indicates an abstainer, a score of 1-7 suggests low-risk consumption, a scores of 8-14 suggest hazardous consumption and a score >15 indicates the likelihood of alcohol dependence.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Prado, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No